CLINICAL TRIAL: NCT05194800
Title: Virtual Mirror Therapy for Relief of Chronic Phantom Limb Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Tech software issues. Unable to complete development
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Conley Carr, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300007560
Record Dates: First submitted 2021-12-06; First posted 2022-01-18 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Phantom Limb Pain
Keywords: Virtual Mirror Therapy; Chronic Phantom Limb Pain
MeSH Terms: conditions — Phantom Limb

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Unilateral upper extremity amputees (Experimental): Unilateral upper extremity amputees suffering from chronic phantom limb pain > 1 yr will be recruited from a hospital based outpatient Physical Medicine and Rehabilitation Amputee Clinic at UAB.
  Interventions: Other: Virtual Mirror Therapy

INTERVENTIONS:
Other: Virtual Mirror Therapy — Subjects will be offered the use of a Virtual Reality headset therapy game. Fiducial markers will be placed on the residual limb for tracking via front facing cameras on the Oculus Quest 2 and the sound limb movements will be duplicated (flipped for chirality) and mapped onto the residual limb to provide the appearance of their residual limb. The software will direct the subjects through a series of guided movements, stretches, and visualization exercises which last a total of 15 minutes. Afterwards the subjects will be given 5 minutes of unstructured time in the program to perform any of exercises or movements they desire in order to attempt to relieve their phantom limb pain.

SUMMARY:
The purpose of this project is to further investigate the use of Virtual Mirror therapy for alleviating symptoms of chronic phantom limb pain. This initial pilot study will inform a fully powered randomized control trial which will include both upper and lower extremity amputees

DETAILED DESCRIPTION:
Ten unilateral upper extremity amputees suffering from chronic phantom limb pain > 1 yr will be recruited from a hospital based outpatient Physical Medicine and Rehabilitation Amputee Clinic. There will be no control group and all 10 subjects will be offered the use of a Virtual Reality headset therapy game (developed in Unreal Engine using Oculus Quest 2 SDK). Fiducial markers will be placed on the residual limb for tracking via front facing cameras on the Oculus Quest 2 and the sound limb movements will be duplicated (flipped for chirality) and mapped onto the residual limb to provide the appearance of their residual limb. The software will direct the subjects through a series of guided movements, stretches, and visualization exercises which last a total of 15 minutes. Afterwards the subjects will be given 5 minutes of unstructured time in the program to perform any of exercises or movements they desire in order to attempt to relieve their phantom limb pain. Subjects will aim for 1 session per week for a total of 6 weeks. Subjects will rate their phantom limb pain symptoms on the Numeric Rating Scale (NRS) prior to and after each session. Prior to the first session as well as at 6 weeks and 12 weeks subjects will rate their phantom limb pain symptoms on the Pain Disability

ELIGIBILITY:
Inclusion Criteria:

* Presence of unilateral upper extremity amputation with continued intermittent or persistent phantom limb pain symptoms > 1 yr after amputation, pain must be >=4 of 10 on the VAS at least intermittently (i.e. can have no pain at times but they must at least have 4/10 intensity of pain when pain does occur).

Exclusion Criteria:

* Uncontrolled bipolar/schizophrenia, active psychosis, uncontrolled seizure disorder, history of severe simulator sickness, active nausea/vomiting, uncontrolled vertigo, bilateral blindness, any facial wounds around the cheeks nose or eyes that may interfere with headset, conjunctivitis, zoster ophthalmicus, immunodeficiency (uncontrolled HIV, immuno-suppressive medications, chemotherapy, etc), severe claustrophobia.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Baseline Numeric Rating Scale of Chronic Phantom Limb Pain | Baseline (Week 0)
  Subjects will rate their phantom limb pain symptoms on the Numeric Rating Scale (NRS) at Baseline to use as comparison to each study session. If pain is intermittent or constant will be noted and if episodic/intermittent a frequency for how often the pain occurs will be obtained as well.
Change from Baseline Numeric Rating Scale at Session1 | Week 1 - Week 52
  Subjects will rate their phantom limb pain symptoms on the Numeric Rating Scale (NRS) prior to and after each session. If pain is intermittent or constant will be noted and if episodic/intermittent a frequency for how often the pain occurs will be obtained as well as if the pain is improved, unchanged, or worsened compared to baseline (prior to study).
Change from Baseline Numeric Rating Scale at Session 2 | Week 2 - Week 52
  Subjects will rate their phantom limb pain symptoms on the Numeric Rating Scale (NRS) prior to and after each session. If pain is intermittent or constant will be noted and if episodic/intermittent a frequency for how often the pain occurs will be obtained as well as if the pain is improved, unchanged, or worsened compared to baseline (prior to study).
Change from Baseline Numeric Rating Scale at Session 3 | Week 3 - Week 52
  Subjects will rate their phantom limb pain symptoms on the Numeric Rating Scale (NRS) prior to and after each session. If pain is intermittent or constant will be noted and if episodic/intermittent a frequency for how often the pain occurs will be obtained as well as if the pain is improved, unchanged, or worsened compared to baseline (prior to study).
Change from Baseline Numeric Rating Scale at Session 4 | Week 4 - Week 52
  Subjects will rate their phantom limb pain symptoms on the Numeric Rating Scale (NRS) prior to and after each session. If pain is intermittent or constant will be noted and if episodic/intermittent a frequency for how often the pain occurs will be obtained as well as if the pain is improved, unchanged, or worsened compared to baseline (prior to study).
Change from Baseline Numeric Rating Scale at Session 5 | Week 5 - Week 52
  Subjects will rate their phantom limb pain symptoms on the Numeric Rating Scale (NRS) prior to and after each session. If pain is intermittent or constant will be noted and if episodic/intermittent a frequency for how often the pain occurs will be obtained as well as if the pain is improved, unchanged, or worsened compared to baseline (prior to study).
Change from Baseline Numeric Rating Scale at Session 6 | Week 6 - Week 52
  Subjects will rate their phantom limb pain symptoms on the Numeric Rating Scale (NRS) prior to and after each session. If pain is intermittent or constant will be noted and if episodic/intermittent a frequency for how often the pain occurs will be obtained as well as if the pain is improved, unchanged, or worsened compared to baseline (prior to study).
Baseline Pain Disability Questionnaire of Chronic Phantom Limb Pain | Baseline (Week 0)
  Prior to the first session as well as at 6 weeks and 12 weeks subjects will rate their phantom limb pain symptoms on the Pain Disability Questionnaire (PDQ).
Change from Baseline Pain Disability Questionnaire at Week 6 | 6 weeks after final session (Session 6)
  Prior to the first session as well as at 6 weeks and 12 weeks subjects will rate their phantom limb pain symptoms on the Pain Disability Questionnaire (PDQ).
Change from Baseline Pain Disability Questionnaire at Week 12 | 12 weeks after final session (Session 6)
  Prior to the first session as well as at 6 weeks and 12 weeks subjects will rate their phantom limb pain symptoms on the Pain Disability Questionnaire (PDQ).

SECONDARY OUTCOMES:
Change in Quality from Baseline Chronic Phantom Limb Pain at Session1 | Week 1 - Week 52
  Free-text section where participants can further describe any changes regarding their pain (change in quality etc).
Change in Quality from Baseline Chronic Phantom Limb Pain at Session 2 | Week 2 - Week 52
  Free-text section where participants can further describe any changes regarding their pain (change in quality etc).
Change in Quality from Baseline Chronic Phantom Limb Pain at Session 3 | Week 3 - Week 52
  Free-text section where participants can further describe any changes regarding their pain (change in quality etc).
Change in Quality from Baseline Chronic Phantom Limb Pain at Session 4 | Week 4 - Week 52
  Free-text section where participants can further describe any changes regarding their pain (change in quality etc).
Change in Quality from Baseline Chronic Phantom Limb Pain at Session 5 | Week 5 - Week 52
  Free-text section where participants can further describe any changes regarding their pain (change in quality etc).
Change in Quality from Baseline Chronic Phantom Limb Pain at Session 6 | Week 6 - Week 52
  Free-text section where participants can further describe any changes regarding their pain (change in quality etc).
Impressions of change from Baseline Chronic Phantom Limb Pain at Session 6 | Week 6 - Week 52
  At the end of 6 sessions of Virtual Mirror Therapy subjects will be given the opportunity to submit opinions/comments regarding their impressions of the sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Conley Carr, MD, Principal Investigator — The University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: No